CLINICAL TRIAL: NCT07209748
Title: The Significance of Soluble CD163 as a Novel Biomarker in the Early Detection and Severity Assessment of HELLP Syndrome
Brief Title: sCD163 in HELLP Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Ragab Hamed Arafa, Principle investigator, Assiut University
Other Study IDs: sCD163 in HELLP syndrome
Record Dates: First submitted 2025-09-30; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: HELLP Syndrome Complicating Pregnancy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control group
  Interventions: Diagnostic Test: sCD163 level
- HELLP Syndrome group
  Interventions: Diagnostic Test: sCD163 level

INTERVENTIONS:
Diagnostic Test: sCD163 level — The significance of soluble CD163 level in the early detection and severity assessment of HELLP Syndrome

SUMMARY:
Primary Aim:

_To investigate the diagnostic potential of soluble CD163 (sCD163)as a novel biomarker for the early detection of HELLP syndrome, assessing its sensitivity and specificity compared to current diagnostic markers.

Secondary Aims:

1. To evaluate the correlation between sCD163 levels and the clinical severity of HELLP syndrome, including complications such as liver dysfunction, thrombocytopenia, and hemolysis.
2. To compare sCD163 levels across different stages of HELLP syndrome (partial vs. complete and other hypertensive disorders of pregnancy (e.g., preeclampsia).

DETAILED DESCRIPTION:
_HELLP syndrome, also known as the syndrome of hemolysis, elevated liver enzymes, and low platelets, represents a sever pregnancy complication typically associated with hypertension. HELLP occurs in 0.2-0.8% of pregnancies and in 70-80% of cases, it coexists with preeclampsia (PE) with a 0-24% mortality rate .Both conditions are classified as hypertensive diseases of pregnancy (HDP), and their pathogenesis has been linked to an excessive maternal inflammatory response, accompanied by enhanced endothelial activation. Erythrocytes are damaged as they pass through blood vessels with impaired endothelium and fibrin strands, resulting in microangiopathic hemolytic anemia (MAHA). Lactate dehydrogenase (LDH) concentration may rise as a consequence of hemolysis. Free hemoglobin binds to unconjugated bilirubin in the spleen or haptoglobin in plasma. Low serum haptoglobin is a characteristic in HELLP women. Patients whose pregnancies are complicated by HELLP syndrome are at a higher risk for renal failure, consumptive coagulopathy, placental abruption, pulmonary and cerebral edema, subcapsular liver hematoma, and hypovolemic shock. Maternal-fetal inflammatory responses were another critical theme , demonstrating that maternal inflammation extends to the fetal compartment, as evidenced by elevated uric acid and CRP in neonates of PE mothers predisposing offspring to long-term metabolic and cardiovascular risks. Soluble clusters of differentiation (sCD163) is a marker of activated macrophages, and its role is to modulate inflammatory reactions. sCD163 stands out as a valuable biomarker, commonly correlates the progression or the severity of several pathological conditions with its levels in tissue fluids, serum, or plasma. It's derived from enzymatic cleavage of cd163 enhanced by inflammatory response or oxidative stress. The primary function attributed to sCD163, similar to CD163, is the absorption and elimination of unbound hemoglobin, thereby reducing oxidative damage caused by heme radicals, since free hemoglobin in the blood stream can contribute to oxidative stress and tissue damage. The scavenging function of sCD163 helps to mitigate these effects. It has been demonstrated that sCD163 and immunoglobulin G interact with the free HB in plasma, leading to monocytic endocytosis of the sCD163-Hb-IgG complex via the Fcγ receptor (FcγR).

Several studies reported significant associations between inflammatory biomarkers and the risk of PE correlating with disease severity, systolic blood pressure, and proteinuria. In our study, we will test levels of sCD163 in pregnant women at different degrees of HELLP syndrome to discover their relationship& its role in early detection of the syndrome.

ELIGIBILITY:
Inclusion Criteria:

* HELLP Syndrome Group:

  1. Pregnant women meeting complete HELLP criteria:

     * Hemolysis (LDH >600 U/L + abnormal smear or bilirubin ≥1.2 mg/dL)
     * AST/ALT ≥70 U/L
     * Platelets <100,000/μL
  2. Gestational age (20-42) weeks
* Control Group:

  1. Normotensive pregnant women (BP <140/90 mmHg, no proteinuria).
  2. Gestational age-matched

Exclusion Criteria:

1. Chronic medical conditionsaffecting sCD163 levels:

   * Autoimmune diseases (e.g., lupus, rheumatoid arthritis)
   * Chronic kidney/liver disease
   * Active infections (e.g., HIV, hepatitis)
2. Fetal anomalies or intrauterine fetal demise at diagnosis.
3. Use of immunosuppressive therapies (e.g., corticosteroids beyond standard HELLP management).
4. Incomplete clinical/laboratory data for HELLP classification.
5. Other gestational disease such as gestational DM

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: * HELLP Syndrome Group:
    1. Pregnant women meeting complete HELLP criteria:
       * Hemolysis (LDH >600 U/L + abnormal smear or bilirubin ≥1.2 mg/dL)
       * AST/ALT ≥70 U/L
       * Platelets <100,000/μL
    2. Gestational age (20-42) weeks
  * Control Group:
    1. Normotensive pregnant women (BP <140/90 mmHg, no proteinuria).
    2. Gestational age-matched
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Comparison of sCD163 level in the 2 study groups | baseline
  To investigate the diagnostic potential of soluble CD163 (sCD163)as a novel biomarker for the early detection of HELLP syndrome, assessing its sensitivity and specificity compared to current diagnostic markers and evaluate the correlation between sCD163 levels and the clinical severity of HELLP syndrome

REFERENCES:
- [Background] Petca A, Miron BC, Pacu I, Dumitrascu MC, Mehedintu C, Sandru F, Petca RC, Rotar IC. HELLP Syndrome-Holistic Insight into Pathophysiology. Medicina (Kaunas). 2022 Feb 21;58(2):326. doi: 10.3390/medicina58020326. PMID 35208649
- [Background] Gardikioti A, Venou TM, Gavriilaki E, Vetsiou E, Mavrikou I, Dinas K, Daniilidis A, Vlachaki E. Molecular Advances in Preeclampsia and HELLP Syndrome. Int J Mol Sci. 2022 Mar 31;23(7):3851. doi: 10.3390/ijms23073851. PMID 35409211
- [Background] Vigil-De Gracia P. Pregnancy complicated by pre-eclampsia-eclampsia with HELLP syndrome. Int J Gynaecol Obstet. 2001 Jan;72(1):17-23. doi: 10.1016/s0020-7292(00)00281-2. PMID 11146072
- [Background] Abdeldaem Mohamed RH, Ahmed Ali Alfaki NM, Belal RE, Ali Dawelbait AM, Hamad Yousif RB, Mohamed SAE, Badre Adam HS, Abbashar Abdelmahmoud EM. Biomarkers of Inflammation and Their Association With the Severity and Onset of Preeclampsia: A Systematic Review. Cureus. 2025 Jul 11;17(7):e87734. doi: 10.7759/cureus.87734. eCollection 2025 Jul. PMID 40786291
- [Background] Plevriti A, Lamprou M, Mourkogianni E, Skoulas N, Giannakopoulou M, Sajib MS, Wang Z, Mattheolabakis G, Chatzigeorgiou A, Marazioti A, Mikelis CM. The Role of Soluble CD163 (sCD163) in Human Physiology and Pathophysiology. Cells. 2024 Oct 11;13(20):1679. doi: 10.3390/cells13201679. PMID 39451197